CLINICAL TRIAL: NCT05804565
Title: Randomised Controlled Trial Comparing Metatarsal Method of Transection Using Bone Cutters or Bone Saw on Outcomes After Ray Amputation (MetaMet)
Brief Title: MetaMet: Bone Cutter Versus Bone Saw for Ray Amputation
Acronym: MetaMet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, Megan Power Foley, Specialist Registrar in Vascular Surgery, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122/12
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot; Gangrene; Limb; Wound Infection; Wound Healing Delayed; Wound Complication; Critical Limb-Threatening Ischaemia; Amputation
Keywords: diabetic foot infection; critical limb ischaemia; minor amputation; reulceration; wound complications
MeSH Terms: conditions — Diabetic Foot; Gangrene; Wound Infection; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: 1:1 parallel randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patient-blinded, assessor-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Saw (Active Comparator): In the "intervention" arm, the metatarsal bone will be transected using an oscillating microsaw. This is an accepted surgical method.
  Interventions: Procedure: Bone Saw
- Bone Cutter (Other): In the "control" arm, the metatarsal bone will be transected using a manual bone cutters. This is also an accepted surgical method
  Interventions: Procedure: Bone Cutter

INTERVENTIONS:
Procedure: Bone Saw — The surgeon will use an oscillating microsaw to transect the metatarsal shaft
  Arms: Bone Saw
Procedure: Bone Cutter — The surgeon will use a manual bone cutter to transect the metatarsal shaft
  Arms: Bone Cutter

SUMMARY:
Toe amputation is a commonly performed operation for infection and/or ischaemia (tissue death due to lack of blood flow). However, a large number of patients having this surgery ultimately require further amputation due to poor wound healing, new infections and/or new ulcers. Research to date has focused on patient-related factors associated with poor wound healing (e.g. diabetes, lack of blood flow, poor kidney function). However, there is no research looking at the technical surgical aspects of the procedure, specifically how the toe bone is cut.

For this feasibility study, we will recruit forty patients whom a consultant vascular surgeon has decided requires amputation of one-to-two adjacent toes. The participants will be randomised by a computer model into one of the two metatarsal transection methods (bone cutters or bone saw) and the rest of the procedure will be carried out in the standard fashion. Patients and assessors will be blinded to which transection method is chosen.

Patients will undergo a post-operative foot x-ray to assess for bone fragments within 48 hours of surgery and another at six months to assess for bone healing. Patients will be asked to rate their pain in the post-operative period using the verbal rating score. Patients will be followed after discharge from hospital by their public health nurse, as is standard practice, with regular follow-up in the surgical outpatients to assess wound progress. Patients will be asked to rate their quality of life at six weeks and six months post-operatively. These assessments will be coordinated with their routine post-operative follow-up clinic appointments, so as not to inconvenience patients with supernumerary visits.

DETAILED DESCRIPTION:
Toe amputation is a common minor vascular procedure and is increasingly performed in the context of irretrievable diabetic foot infection, with and without concurrent ischaemia. Approximately 422 million people worldwide have diabetes mellitus and peripheral arterial disease (PAD) affects approximately 200 million people(1). The intersection between diabetes, neuro-ischaemic foot ulceration and lower limb amputations is well established(2). Recently published data from the United States reported overall rates of lower limb amputations in diabetic patients rose between 2000 and 2015, in part due to a 62% increase in the rate of minor (foot and toe) amputations(3). It is estimated that 6% of Irish adults are diabetic; from this, we can extrapolate the burden of managing diabetic foot complications(4). Resource utilisation notwithstanding, the financial costs of managing diabetic foot complications are estimated to outstrip some cancers(5). As the prevalence of diabetes mellitus rises amongst an ageing Irish population, the importance of achieving durable functional outcomes after partial foot amputation is paramount.

Re-ulceration, re-infection, re-amputation and hospital re-admission after partial foot amputation for digital gangrene is well documented in the literature in both diabetic and PAD cohorts(6). Across the literature, rates of re-amputation at five years post-index surgery for diabetic foot complications range from 45-65% (6, 7). A recent study by Collins et al reported that, out of 146 Irish patients undergoing minor amputations, 43% (n=63) required further ipsilateral amputation, 21 (14.4%) of which were trans-tibial or trans-femoral(8). Chronic kidney disease, diabetes with or without poor gylcaemic control, peripheral neuropathy, peripheral arterial disease, ongoing tobacco smoking, obesity (BMI >30), concurrent sepsis at the time of index operation have all been identified as independent risk factors for amputation failure and the need for revision(9-11). While numerous studies have investigated patient-dependent factors predictive of amputation failure, there is a dearth of evidence examining the impact of surgical technique on this commonly performed procedure.

An exhaustive search of the literature surrounding surgical technique and outcomes after ray amputation yielded several papers on the benefits of various soft tissue flaps for covering wound defects but just one detailing a particular methods of bone transection. However, Moodley et al focused on the use of a Gigli saw, which is beyond the scope of this feasibility study(12). There have been no randomised controlled trials evaluating the impact of metatarsal transection method on outcomes after ray amputation, specifically whether a manual bone cutter or an electric/oscillating/pneumatic bone saw were used. We hypothesise that utilising a manual bone cutter is more subject to inter-user variability, as it depends on the physical strength of the operating surgeon; improperly applied forces are liable to fracture the remaining bone, leaving small comminuted fragments that may become necrotic and act as a nidus for further infection within the wound bed. Furthermore, using an oscillating microsaw has the advantage of providing a clean bony transection regardless of the physical strength of the operator, however it may cause more damage to the surrounding connective tissues and disturb microvascular periosteal supply, which could also lead to osteonecrosis. We propose a pilot randomised controlled trial to test the feasibility and to generate sufficient data to permit sample size calculation for a trial designed to evaluate the outcomes after ray amputation using either a bone cutter or a bone saw.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients, aged 18 and over, undergoing transmetatarsal amputation of one-to-two adjacent toes

Exclusion Criteria:

* Significant peripheral arterial disease, as defined by ABPI <0.4 or digital pressures of <50mmHg, not undergoing concurrent revascularisation;
* Patients undergoing amputation of three of more adjacent toes
* Patients unfit for surgery;
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Power Calculation for Definitive RTC | Six months
  collect sufficient data to enable an accurate power calculation for a future randomised controlled trial

SECONDARY OUTCOMES:
Rate of Surgical Re-Intervention | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on rates of surgical reintervention at the index procedure site
Rate of Hospital Re-Admissions | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on rates of hospital re-admissions directly related to the index surgical procedure
Time to Wound Healing | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on time to healing of the index surgical wound
Rate of Index Ulcer Healing | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on healing of the index ulcer
Rate of Re-Infection | six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on rates of re-infection at the index procedure site
Rate of Ulcer Recurrence | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on ulcer recurrence or further ulceration
Rate of Recurrent Osteomyelitis | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on osteomyelitis recurrence adjacent to the index surgical site
Rate of Resection Margin Positive Culture | Six months
  To determine the effect of microsaw compared to bone cutters for toe amputation on resection margin culture positivity
Patient-Reported Post-Operation Pain | Six Months
  To determine the effect of microsaw compared to bone cutters for toe amputation on patient-reported post-operative pain, as measured by the Verbal Rating Scale (VRS)
Patient-Reported Quality of Life | Six Months
  To determine the effect of microsaw compared to bone cutters for toe amputation on patient-reported health-related quality of life at six weeks and six months, as measured by the EQ-5D-5L tool

CONTACTS AND LOCATIONS:
Overall Officials: Stewart R Walsh, FRCS, Principal Investigator — University College Hospital Galway
Locations (1):
- University College Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shu J, Santulli G. Update on peripheral artery disease: Epidemiology and evidence-based facts. Atherosclerosis. 2018 Aug;275:379-381. doi: 10.1016/j.atherosclerosis.2018.05.033. Epub 2018 May 22. No abstract available. PMID 29843915
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] Geiss LS, Li Y, Hora I, Albright A, Rolka D, Gregg EW. Resurgence of Diabetes-Related Nontraumatic Lower-Extremity Amputation in the Young and Middle-Aged Adult U.S. Population. Diabetes Care. 2019 Jan;42(1):50-54. doi: 10.2337/dc18-1380. Epub 2018 Nov 8. PMID 30409811
- [Background] Nolan JJ, O'Halloran D, McKenna TJ, Firth R, Redmond S. The cost of treating type 2 diabetes (CODEIRE). Ir Med J. 2006 Nov-Dec;99(10):307-10. PMID 17274175
- [Background] Skrepnek GH, Mills JL Sr, Lavery LA, Armstrong DG. Health Care Service and Outcomes Among an Estimated 6.7 Million Ambulatory Care Diabetic Foot Cases in the U.S. Diabetes Care. 2017 Jul;40(7):936-942. doi: 10.2337/dc16-2189. Epub 2017 May 11. PMID 28495903
- [Background] Armstrong DG, Lavery LA, Harkless LB, Van Houtum WH. Amputation and reamputation of the diabetic foot. J Am Podiatr Med Assoc. 1997 Jun;87(6):255-9. doi: 10.7547/87507315-87-6-255. PMID 9198345
- [Background] Rathnayake A, Saboo A, Malabu UH, Falhammar H. Lower extremity amputations and long-term outcomes in diabetic foot ulcers: A systematic review. World J Diabetes. 2020 Sep 15;11(9):391-399. doi: 10.4239/wjd.v11.i9.391. PMID 32994867
- [Background] Collins PM, Joyce DP, O'Beirn ES, Elkady R, Boyle E, Egan B, Tierney S. Re-amputation and survival following toe amputation: outcome data from a tertiary referral centre. Ir J Med Sci. 2022 Jun;191(3):1193-1199. doi: 10.1007/s11845-021-02682-4. Epub 2021 Jun 22. PMID 34156661
- [Background] Acar E, Kacira BK. Predictors of Lower Extremity Amputation and Reamputation Associated With the Diabetic Foot. J Foot Ankle Surg. 2017 Nov-Dec;56(6):1218-1222. doi: 10.1053/j.jfas.2017.06.004. Epub 2017 Jul 29. PMID 28765052
- [Background] Liu R, Petersen BJ, Rothenberg GM, Armstrong DG. Lower extremity reamputation in people with diabetes: a systematic review and meta-analysis. BMJ Open Diabetes Res Care. 2021 Jun;9(1):e002325. doi: 10.1136/bmjdrc-2021-002325. PMID 34112651
- [Background] Norvell DC, Czerniecki JM. Risks and Risk Factors for Ipsilateral Re-Amputation in the First Year Following First Major Unilateral Dysvascular Amputation. Eur J Vasc Endovasc Surg. 2020 Oct;60(4):614-621. doi: 10.1016/j.ejvs.2020.06.026. Epub 2020 Aug 13. PMID 32800475
- [Background] Moodley B, Grabowski G, Altschuler M, Williams M. Use of the Gigli saw for transmetatarsal amputations. J Foot Ankle Surg. 2005 Sep-Oct;44(5):415-8. doi: 10.1053/j.jfas.2005.07.013. No abstract available. PMID 16210164

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05804565/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05804565/ICF_001.pdf